CLINICAL TRIAL: NCT01088464
Title: A Phase 1 Study of IMC-11F8 in Patients With Advanced Solid Tumors
Brief Title: Study of IMC-11F8 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13904; CP11-0907 (Other: ImClone Systems); I4X-IE-JFCA (Other: Eli Lilly); 21-1901 (Other: PMDA (MoH) in Japan)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasms
Keywords: Human Immunoglobulin Gamma-1 (IgG1); Monoclonal Antibody (MAb); Epidermal Growth Factor Receptor (EGFR); Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Biological: IMC-11F8
- Cohort 2 (Experimental)
  Interventions: Biological: IMC-11F8
- Cohort 3 (Experimental)
  Interventions: Biological: IMC-11F8

INTERVENTIONS:
Biological: IMC-11F8 — 600 milligrams (mg) intravenously, Days 1 and 8 every 3 weeks
  Other Names: Necitumumab; LY3012211
  Arms: Cohort 1
Biological: IMC-11F8 — 800 mg intravenously, every 2 weeks
  Other Names: Necitumumab; LY3012211
  Arms: Cohort 2
Biological: IMC-11F8 — 800 mg intravenously, Days 1 and 8 every 3 weeks
  Other Names: Necitumumab; LY3012211
  Arms: Cohort 3

SUMMARY:
This study is to establish the safety and pharmacokinetic (PK) profile of IMC-11F8, administered either: (1) in a 3-week cycle; or (2) in a 2-week cycle to Japanese participants with advanced solid tumors who have not responded to standard therapy or for whom no standard therapy is available.

DETAILED DESCRIPTION:
This single center, open-label, single-arm, Phase 1 study will enroll 18 participants at a maximum. The actual size will vary depending on the dose-limiting toxicities (DLTs) observed and the resultant sizes of the cohorts. Participants will receive IMC-11F8 administered intravenously, once every 2 weeks or on Days 1 and 8 every 3 weeks for 6 weeks (1 cycle). All infusions can be administered within ± 1 day of the scheduled administration date. After 1 cycle of treatment, participants who have an objective response or stable disease may continue to receive IMC-11F8 at the same dose and schedule until disease progression or other withdrawal criteria are met.

A minimum of 3 participants will be enrolled in each cohort. Dose escalation in successive cohorts will occur once all participants complete 1 cycle of therapy.

Participants will be enrolled sequentially into each cohort. A completed participant will be either a participant who completes the initial 6-week treatment period (Cycle 1) or a participant who discontinues therapy for an IMC-11F8-related toxicity during Cycle 1. Participants who do not complete the first 6 weeks of treatment for reasons other than an IMC-11F8-related toxicity will be replaced. Toxicity data for each cohort will be reviewed prior to dose escalation. Upon completion of all required safety evaluations during the initial 6 weeks, the next cohort of new participants will be treated at the next higher dose level using a dose escalation scheme.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor participant who has been histopathologically or cytologically documented
* Advanced primary or recurrent solid tumors participant who has not responded to standard therapy or for whom no standard therapy is available
* The participant has measurable or nonmeasurable lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 guidelines
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1 at study entry
* The participant is able to provide written informed consent
* The participant is age 20 years or older
* The participant has a life expectancy of > 3 months
* The participant has adequate hematologic function
* The participant has adequate renal function
* The participant agrees to use adequate contraception for the duration of study participation and for at least 12 weeks after the last dose of study therapy
* The participant has adequate recovery from recent surgery, chemotherapy, and radiation therapy (including palliative radiation therapy). At least 28 days (6 weeks for nitrosoureas or mitomycin C) must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy. For treatment with nonapproved monoclonal antibodies, a minimum of 8 weeks must have elapsed
* The participant is willing to comply with study procedures until the End-of-Therapy visit

Exclusion Criteria:

* The participant has received chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or the participant has ongoing side effects ≥Grade 2 due to agents administered more than 28 days earlier (except alopecia)
* The participant has documented and/or symptomatic brain or leptomeningeal metastases (participants who are clinically stable [no symptoms during the 4 weeks prior to enrollment] with an assessment that no further treatment [radiation, surgical excision, or administration of steroids] is required are permitted to enter the study)
* The participant has an uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic antibiotic treatment
  * Congestive heart failure (Class III or IV per the New York Heart Association heart disease classification guidelines)
* The participant has participated in clinical studies of nonapproved experimental agents or procedures within 4 weeks prior to first dose of study therapy, or within 8 weeks prior to first dose of study therapy for nonapproved monoclonal antibodies
* The participant has received any previous treatment with monoclonal antibodies targeting the epidermal growth factor receptor (EGFR). Previous treatment with EGFR tyrosine kinase inhibitors (TKI), approved or nonapproved, is allowed. There must be a time interval of at least 4 weeks between the last EGFR TKI dose and the first dose of IMC-11F8
* The participant has acute or subacute intestinal occlusion/obstruction
* The participant has a history of inflammatory bowel disease (for example, Crohn's disease, ulcerative colitis) requiring medical intervention in the 3 years prior to study entry
* The participant has acute pulmonary disorder, interstitial pneumonia, pulmonary fibrosis, or history thereof
* The participant has a known allergy to any of the treatment components, or to monoclonal antibodies or other therapeutic proteins such as fresh frozen plasma, human serum albumin, cytokines, or interleukins. In the event that there is suspicion that the participant may have allergies, the participant should be excluded
* The participant, if female, is pregnant (confirmed by urine or serum pregnancy test) or lactating
* The participant has known alcohol or drug dependency
* The participant is hepatitis B virus (HBV) antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody positive
* The participant is assessed as inadequate for the study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had 3 cohorts and dose escalation in successive cohorts was to occur once all the participants completed 1 cycle of therapy. A completed participant was either a participant who completed the initial 6-week treatment period (Cycle 1) or a participant who discontinued therapy for an IMC-11F8 (Necitumumab) related toxicity during Cycle 1.
Groups:
- Cohort 1: Necitumumab: Necitumumab 600 milligrams (mg) administered intravenously on Days 1 and 8 every 3 weeks of a 6-week cycle. After Cycle 1, participants showing objective response or stable disease were to receive necitumumab at same dose and schedule until disease progression or other withdrawal criteria were met.
- Cohort 2: Necitumumab: Necitumumab 800 mg administered intravenously every 2 weeks of a 6-week cycle. After Cycle 1, participants showing objective response or stable disease were to receive necitumumab at same dose and schedule until disease progression or other withdrawal criteria were met.
- Cohort 3: Necitumumab: Necitumumab 800 mg administered intravenously on Days 1 and 8 every 3 weeks of a 6-week cycle. After Cycle 1, participants showing objective response or stable disease were to receive necitumumab at same dose and schedule until disease progression or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Started | 3 | 6 | 6
Received Any Quantity of Study Drug | 3 | 6 | 6
Completed | 3 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received any quantity of study drug.
Groups:
- Cohort 1: Necitumumab: Necitumumab 600 mg administered intravenously on Days 1 and 8 every 3 weeks of a 6-week cycle. After Cycle 1, participants showing objective response or stable disease were to receive necitumumab at same dose and schedule until disease progression or other withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15
Age, Continuous [Median (Full Range); unit: years] | 57.2 (20.02) [30.5 to 69.6] | 64.5 (4.51) [56.2 to 68.9] | 56.7 (9.50) [51.3 to 75.6] | 61.2 (10.72) [30.5 to 75.6]
Gender [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 2 | 3 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 3 | 6 | 6 | 15
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 6 | 6 | 15
Eastern Cooperative Oncology Group performance status (ECOG PS) [Number; unit: participants] — ECOG PS was used to classify participants according to their functional impairment. Score 0 = Fully active, able to carry on all pre-disease performance without restriction. Score 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, for example, light house work, office work.
  participants
    0 = Fully Active | 1 | 1 | 4 | 6
    1 = Ambulatory, Restricted Work Activity | 2 | 5 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: Data presented are the number of participants who experienced 1 or more TEAEs or SAEs regardless of causality. An adverse event was considered as TEAE if it occurred any time after the administration of the first dose of study drug or up to 30 days after the last dose of study treatment or if it occurred prior to the first dose and worsened while on treatment. A summary of SAEs and other non-SAEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to 24 weeks plus 30 days post last dose of study drug
Population: All participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
participants
  TEAEs | 3 | 6 | 6
  SAEs | 1 | 0 | 1

2. Primary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of Necitumumab After a Single Dose
Time Frame: Cycle 1, Day 1; Cohorts 1 and 3: predose, immediately after end of infusion, 0.5, 1, 2, 6, 24, 96 and 168 hours (h) after end of infusion. Cohort 2: predose, immediately after infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 h after end of infusion
Population: All participants who received single dose of study drug and had Cmax values for Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
micrograms per milliliter (µg/mL) | 306 (29) | 417 (46) | 352 (20)

3. Primary Outcome: PK: Cmax of Necitumumab After Multiple Doses
Description: Cmax at steady state (after the last dose of the initial 6-week treatment cycle).
Time Frame: Cycle 1, Day 29; For Cohorts 1, 2 and 3: predose (prior to fourth infusion for Cohorts 1 and 3; prior to third infusion for Cohort 2), immediately after end of infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 h after end of infusion
Population: All participants who received multiple doses of study drug and had Cmax values for Day 29 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
µg/mL | 396 (5) | 523 (17) | 629 (16)

4. Primary Outcome: PK: Minimum Concentration (Cmin) of Necitumumab After a Single Dose
Description: Cmin is defined as the minimum concentration the drug achieved after administration of first infusion and prior to the administration of second infusion.
Time Frame: Cycle 1; Cohorts 1, 2 and 3: prior to second infusion
Population: All participants who received single dose of study drug and had Cmin serum concentrations analyzed prior to administration of second dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
µg/mL | 86.0 (10) | 72.9 (24) | 127 (18)

5. Primary Outcome: PK: Cmin of Necitumumab After Multiple Doses
Description: Cmin was calculated prior to the last dose of the initial 6-week treatment cycle.
Time Frame: Cycle 1; Cohorts 1and 3: prior to fourth infusion. Cohort 2: prior to third infusion
Population: All participants who received multiple doses of study drug and had Cmin serum concentrations prior to last dose of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 5
µg/mL | 108 (23) | 136 (22) | 220 (16)

6. Primary Outcome: PK: Area Under the Concentration-Time Curve From Time 0 to Last Time Point [AUC (0-tlast)] of Necitumumab After a Single Dose
Time Frame: Cycle 1, Day 1; Cohorts 1 and 3: predose, immediately after end of infusion, 0.5, 1, 2, 6, 24, 96 and 168 h after end of infusion. Cohort 2: predose, immediately after end of infusion, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264 and 336 h after end of infusion
Population: All participants who received single dose of study drug and had evaluable AUC(0-∞) values for Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*h/mL)
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
micrograms*hour/milliliter (µg*h/mL) | 23100 (16) | 50100 (24) | 31300 (17)

7. Primary Outcome: PK: Area Under the Concentration-Time Curve From Time 0 to Infinity [AUC(0-∞)] of Necitumumab After a Single Dose
Description: AUC(0-∞) was calculated only for participants in Cohort 2 as the percentage of AUC extrapolated beyond tlast was greater than 30% for all the remaining participants.
Time Frame: as for outcome 6
Population: All participants who received single dose of study drug and had evaluable AUC(0-∞) values for Day
  1 of Cycle 1. No participant of Cohorts 1 and 3 were analyzed for AUC(0-∞) on Day 1 of Cycle 1, due to fraction of data outside tlast >30%
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 0 | 3 | 0
µg*h/mL |  | 66700 (21) |

8. Secondary Outcome: Immunogenicity (IK): Number of Participants With Treatment-Emergent Anti-IMC-11F8 Antibodies
Description: Treatment-emergent samples were defined as samples which showed at least 4-fold difference (2 dilution increase) at post-baseline in IK titer over the baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20).
Time Frame: For Cohorts 1, 2 and 3: Prior to first infusions of Cycles 1, 2, and 4 and at the 30-day follow-up visit (+7 days) after the last dose of study drug
Population: All participants who received any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
participants
  Positive for Anti-Necitumumab Antibodies | 0 | 0 | 0
  Negative for Anti-Necitumumab Antibodies | 3 | 6 | 6

9. Primary Outcome: PK: Area Under the Concentration-Time Curve From Time 0 to 336 h Postdose [AUC(0-336)] of Necitumumab After Multiple Doses
Description: Steady state AUC(0-336) values are reported.
Time Frame: as for outcome 3
Population: All the participants who received multiple doses of study drug and had AUC(0-336) values for Day 29 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 5
µg*h/mL | 56300 (21) | 81400 (19) | 105000 (12)

10. Primary Outcome: PK: Half-Life (t½) of Necitumumab After a Single Dose
Description: The t½ is defined as the time taken for study drug in blood to decrease to half of its concentration.
Time Frame: as for outcome 6
Population: All participants who received single dose of study drug and had t½ values for Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 6 | 6
h | 126 (14) | 207 (31) | 146 (18)

11. Primary Outcome: PK: t½ of Necitumumab After Multiple Doses
Description: The t½ is defined as the time taken for study drug in blood to decrease to half of its concentration.
Time Frame: as for outcome 3
Population: All the participants who received multiple doses of study drug and had t½ values for Day 29 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 3 | 5 | 5
h | 190 (36) | 233 (18) | 286 (18)

12. Primary Outcome: PK: Clearance (CL) of Necitumumab After a Single Dose
Description: CL is defined as the volume of plasma that is cleared of study drug per unit time. CL was not analyzed for participants in Cohorts 1 and 3 as CL is derived from AUC(0-∞). AUC(0-∞) was calculated only for participants in Cohort 2 as the percentage of AUC extrapolated beyond tlast was greater than 30% for the remaining participants.
Time Frame: as for outcome 6
Population: All the participants who received single dose of study drug and had CL values for Day 1 of Cycle 1. No participant of Cohorts 1 and 3 were analyzed for CL on Day 1 of Cycle 1, due to fraction of data outside tlast >30%
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour (mL/h)
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 0 | 3 | 0
milliliters per hour (mL/h) |  | 12.0 (21) |

13. Primary Outcome: PK: CL of Necitumumab After Multiple Doses
Description: CL is defined as the volume of plasma that is cleared of study drug per unit time. Data did not allow calculation of CL for participants in Cohorts 1 and 3.
Time Frame: as for outcome 3
Population: All the participants who received multiple doses of study drug and had CL values for Day 29 of Cycle 1. CL of necitumumab was not assessed for participants in Cohorts 1 and 3, due to the irregular dosing regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 0 | 6 | 0
mL/h |  | 9.83 (19) |

14. Primary Outcome: PK: Steady-State Volume of Distribution (Vss) of Necitumumab After Single Dose
Description: Vss is that amount of plasma in which the study drug needs to be dissolved to attain a steady state drug concentration. Vss was not analyzed for participants in Cohorts 1 and 3 as Vss is derived from AUC (0-∞). AUC(0-∞) was calculated only for participants in Cohort 2 as the percentage of AUC extrapolated beyond tlast was greater than 30% for the remaining participants.
Time Frame: as for outcome 6
Population: All participants who received single dose of study drug and had Vss values for Day 1 of Cycle 1. Vss of necitumumab was not assessed for participants in Cohorts 1 and 3, due to the irregular dosing regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters (mL)
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 0 | 3 | 0
milliliters (mL) |  | 2780 (31) |

15. Primary Outcome: PK: Vss of Necitumumab After Multiple Doses
Description: Vss is that amount of plasma in which the study drug needs to be dissolved to attain a steady state drug concentration. Data did not allow calculation of Vss for participants in Cohorts 1 and 3.
Time Frame: as for outcome 3
Population: All participants who received multiple doses of study drug and had Vss values for Day 29 of Cycle 1. Vss of necitumumab was not assessed for participants in Cohorts 1 and 3, due to the irregular dosing regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Number analyzed (Participants) | 0 | 5 | 0
mL |  | 3370 (21) |

ADVERSE EVENTS:
Time Frame: Baseline up to 24 weeks plus 30 days post last dose of study drug
Arm/Group | Cohort 1: Necitumumab | Cohort 2: Necitumumab | Cohort 3: Necitumumab
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Necitumumab (N=3) | Cohort 2: Necitumumab (N=6) | Cohort 3: Necitumumab (N=6)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Necitumumab (N=3) | Cohort 2: Necitumumab (N=6) | Cohort 3: Necitumumab (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (4) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (4) | 3 (3)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (6) | 4 (4)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 5 (8)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (7) | 2 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 2 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study completion or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.